CLINICAL TRIAL: NCT07402317
Title: Outcome of a New Trimodality Bladder Perservation Protocol for Patients With Muscle Invasive Bladder Cancer
Brief Title: Trimodality Bladder Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Esmail Ali Abdelbaki, Assistant lecturer, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bladder cancer treatment
Record Dates: First submitted 2026-02-01; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T2 bladder cancer (Experimental): T2 patients
  Interventions: Procedure: Transurethral resection of bladder tumor: We are aimed at Complete TURBT. Which was defined as no residual tumor, whereas incomplete TURBT

INTERVENTIONS:
Procedure: Transurethral resection of bladder tumor: We are aimed at Complete TURBT. Which was defined as no residual tumor, whereas incomplete TURBT — Neo adjuvant chemotherapy followed by turbt followed by radiotherapy

SUMMARY:
The aim of this study is To evaluate the outcomes of patients with muscle invasive bladder cancer managed by trimodal therapy", Neoadjuvant chemotherapy( NAC) followed by Transurethral resection of the bladder tumor then Radiotherapy, for bladder preservation and capability to reach the goal of better quality of life, compared to radical cystectomy with assessment of factors that may predict treatment response, risk of recurrences and (disease- free and over all)survival of such patients...

DETAILED DESCRIPTION:
Bladder Cancer (BC) is a worldwide health problem. It is the 7th most commonly diagnosed cancer in male population worldwide, whilst it drops to 11th for both sexes. Approximately 25% of newly diagnosed patients have muscle-invasive disease. Despite potentially curative radical surgery, approximately 50% of muscle invasive cases develop relapse within 2 years, and most of them die. Organ preservation has been the main goal of cancer care in the last two decades, yet it is not generally adopted for the cure of non-metastatic muscle invasive bladder cancer[1].

The standard of care for muscle invasive urothelial-cell carcinoma (UCC) of the bladder is radical cystectomy (RC). Radical surgery results in long-term survival rates of 40%-60% [2-4]. Sophisticated techniques for urinary diversion have been developed to improve patients' quality of life; however, this cannot substitute for the patient's original bladder [5].

Attempts to obtain bladder preservation are only justified when they have a high likelihood of achieving local cure with no compromise in survival rates. Transurethral resection of the bladder tumor (TURBT) alone, chemotherapy alone or radiation therapy alone provide inferior outcomes to radical cystectomy with only 20% to 40% local control rates in muscle invasive urothelial-cell carcinoma (UCC). Several groups have reported the value of combining all three modalities, with salvage cystectomy being reserved for patients with incomplete response or local relapse [6,7]. Bladder preservation approaches became increasingly favored, and became successful , essentially after the emergence of concurrent chemo-radiation protocols with cisplatin. The National Bladder Cancer Group first demonstrated the safety and efficacy of cisplatin, as a radiation sensitizer, in patients with MIBC who were unsuitable for cystectomy[8].

ELIGIBILITY:
Inclusion Criteria: clinical case's of muscle invasive bladder cancer .T2 or more bladder cancer according to the American Joint Committee on Cancer (AJCC) staging system.

* Age >18 years old. .Adequate bone marrow function. .Adequate renal functions. .Adequate hepatic functions.

Exclusion criteria:

.Distant metastases, pelvic lymph node metastasis. .Evidence of tumor-related hydronephrosis. .Severe irritative bladder symptoms.

* Persistent infection. .Associated serious medical or psychiatric illness. .Prior or concurrent malignancy of any other site unless the patient was disease free for 5 years.

.Previous systemic chemotherapy or pelvic irradiation. .Pregnant or lactating female patients. .Each patient will give written informed consent before entering the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Clinical ,radiological response , diagnostic cystoscopy and turbt biopsy either before and after neo adjuvant chemotherapy. Assessed response either complete, partial or progressive . according to tumor size,site ,stage, biopsy ( complete or incomplete | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Azhar Assiut faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] https://pubmed.ncbi.nlm.nih.gov/23485231/
- See also: Pub med — https://pubmed.ncbi.nlm.nih.gov/23485231/